CLINICAL TRIAL: NCT03975569
Title: Studie Van de Vaginale Microbiota en Het Potentieel Van Een Vaginale Zalf Met Probiotica Bij Vaginale Candidose
Brief Title: Study of the Vaginal Microbiota and the Potential of a Vaginal Probiotic Cream in Vaginal Candidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Ethisch Comité, UZA, Prof. Dr. Gilbert Donders, MD, PhD, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16/7/66; B300201628296 (Other: Belgian Registration)
Record Dates: First submitted 2019-02-12; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Candidiasis, Vulvovaginal
Keywords: vaginal, yeast infection, candida, candidosis
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Torulopsis; Candidiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vulvovaginitis patients- lactobacillus gel (Experimental): Daily use of vaginal gel containing lactobacilli by patients. Probiotic vaginal gel.
  Interventions: Other: Probiotic vaginal gel

INTERVENTIONS:
Other: Probiotic vaginal gel — Total daily administration of 2.5 ml of probiotic gel, containing three lactobacilli (Lactobacillus rhamnosus GG, Lactobacillus pentosus KCA1 and Lactobacillus plantarum WCFS1). Final dosage per gram of gel: 10^9-10^10 colony forming units of lactobacilli.

SUMMARY:
This study evaluated the effect of a vaginal gel containing three live probiotic bacteria on vaginal Candida albicans infection in flemish patients (n=20). The therapeutic effects of the gel will be clinically evaluated (vaginal pH, microscopic and clinical scores). The effect on the vaginal microbiome will be evaluated through 16S ribosomal RNA amplicon sequencing via MiSeq Illumina and polymerase chain reaction (PCR) for Candida albicans.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* willing to adhere to protocol
* premenopausal
* positive Candida microscopy and/or culture
* at least two of the following vaginal symptoms: burning, itching, redness, fissure, discharge, vulvar edema, postcoital itching, lesions with partner

Exclusion Criteria:

* vaginal use of any products 1 week or less before randomization
* use of oral or local antimycotic treatment 1 week or less before randomization
* unprotected sexual contact 24 hours preceding randomization
* vaginal douching 24 hours preceding randomization
* patient does not agree to participate in the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Vaginal persistence of Candida species | through study completion, estimated 1 year
  The presence of Candida species in the collected samples will be analyzed by microscopy, culture (clinical lab) and after DNA extraction through quantitative PCR as molecular method. This will allow to estimate relative and absolute concentrations of the suspected infectious agent, and allow to evaluate if the infection cleared or not.

SECONDARY OUTCOMES:
Clinical scores of patients | through study completion, estimated 1 year
  By the responsible gynecologist, symptom severity (burning, itching, redness, swelling and fissures) was estimated and scored as absent, mild, moderate or severe. This will provide information about the ability of the gel to ameliorate the symptoms of vulvovaginal candidosis.
Microbiome analysis | through study completion, estimated 1 year
  After Illumina MiSeq sequencing, bio-informatics tools will be used to cluster bacteria and yeasts into operation taxonomic units/ amplicon sequence variants (ASVs). Based on these ASVs, the bacterial and fungal community will be compared over the sampled periods and allow comparison of the composition over the study period. The investigators will specifically screen for ASVs that can be expected to be derived from supplied probiotic strains or that are responsible for the infection (expected Candida ASVs). Additionally, the investigators will pay attention to the dominant members of the vaginal bacterial community (expected in most women to be dominated by one of four Lactobacillus species).